CLINICAL TRIAL: NCT01554631
Title: Randomized, Non-blinded, 3-fold Crossover Study to Investigate the Bioequivalence Between Glucobay ODT 100 mg Taken Without and With Water and the Glucobay Standard Tablet 100 mg Following Single Oral Dosing in Healthy Male Subjects
Brief Title: A 3-fold Crossover Bioequivalence Study Between Glucobay ODT (Orally Disintegrating Tablet) 100 mg and Glucobay Standard Tablet 100 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer Healthcare AG
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 16025; 2012-000245-12 (EudraCT Number)
Record Dates: First submitted 2012-03-07; First posted 2012-03-15 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Bioequivalence; Acarbose; ODT
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Day 0: oral sucrose load (75 g sucrose dissolved in 225 mL water) without Glucobay ODT 100 mg; Day 1: oral sucrose load plus Glucobay ODT 100 mg taken without water
  Interventions: Drug: Acarbose (Glucobay ODT, BAYG5421)
- Arm 2 (Experimental): Day 0: oral sucrose load (75 g sucrose dissolved in 225 mL water) without Glucobay ODT 100 mg; Day 1: oral sucrose load plus Glucobay ODT 100 mg taken with water
  Interventions: Drug: Acarbose (Glucobay ODT, BAYG5421)
- Arm 3 (Active Comparator): Day 0: oral sucrose load (75 g sucrose dissolved in 225 mL water) without Glucobay standard tablet 100 mg; Day 1: oral sucrose load plus Glucobay standard tablet 100 mg taken with water
  Interventions: Drug: Acarbose (Glucobay, BAYG5421)

INTERVENTIONS:
Drug: Acarbose (Glucobay ODT, BAYG5421)
  Arms: Arm 1; Arm 2
Drug: Acarbose (Glucobay, BAYG5421)
  Arms: Arm 3

SUMMARY:
To establish the bioequivalence between Glucobay ODT (Orally Disintegrating Tablet) 100 mg taken without or with water and the Glucobay standard tablet 100 mg taken with water.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Age: 18 to 45 years (inclusive) at the first screening examination / visit
* Ethnicity: White
* Body mass index (BMI): above/equal 18 and below/equal 28 kg / m²

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Subjects with a medical disorder, condition or history of such that would impair the subject's ability to participate or complete this study in the opinion of the investigator or the sponsor
* Known hypersensitivity to the study drugs (active substances or excipients of the preparations)
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Chronic intestinal disorders associated with distinct disturbances of digestion and absorption
* States which may deteriorate as a result of increased gas formation in the intestine (e.g. Roemheld´s syndrome, major hernias, intestinal obstructions, intestinal ulcers, Crohn´s disease, ulcerative colitis, malabsorptions)
* Fasting blood glucose level outside normal range
* Impaired glucose tolerance in glucose tolerance test

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Ratio of postprandial maximum concentration (Cmax) of blood glucose following sucrose load with Glucobay (Day 1) and without Glucobay (Day 0) | within 4 hours after sucrose load
Ratio of postprandial Area under curve from 0 to 4 hours (AUC(0-4)) of blood glucose following sucrose load with Glucobay (Day 1) and without Glucobay (Day 0) | within 4 hours after sucrose load

SECONDARY OUTCOMES:
Difference in postprandial maximum concentration (Cmax) of blood glucose and serum insulin following sucrose load with acarbose (day 1) and without acarbose (day 0) | within 4 hours after sucrose load
Difference in postprandial area under curve from 0 to 4 hours (AUC(0-4)) of blood glucose and serum insulin following sucrose load with acarbose (day 1) and without acarbose (day 0) | within 4 hours after sucrose load
Safety parameters | Assessed in pre study treatment, study treatment, and follow-up visits
  Adverse events (AEs), clinical chemistry, hematology, urinalysis, physical examination, systolic and diastolic blood pressure, pulse rate, electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Mönchengladbach, North Rhine-Westphalia, Germany